CLINICAL TRIAL: NCT05051059
Title: Assessment of the Functional Outcome and Quality of Life in Sarcoma Patients
Acronym: QOLSarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S63146
Record Dates: First submitted 2021-09-09; First posted 2021-09-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma
Keywords: Lower extremities; Health related quality of life; Functional outcome; Limb salvage surgery
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Quality of Life; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Soft tissue sarcoma of the thigh (Other): Patients who underwent surgical resection of a deep intramuscular soft tissue sarcoma of the thigh
  Interventions: Other: Functional outcome; Other: Health related quality of life (HRQoL) assessment
- Control group (No Intervention): A group of healthy age-matched individuals will be identified out of an available gait lab database to compare the gait pattern with tha of the patient group
- Bone or soft tissue sarcoma of the lower extremity (Other): Patients who underwent surgical resection of a bone or soft tissue sarcoma of the lower extremity
  Interventions: Other: Health related quality of life (HRQoL) assessment

INTERVENTIONS:
Other: Functional outcome — 3D-motion analysis and strength assessment
  Arms: Soft tissue sarcoma of the thigh
Other: Health related quality of life (HRQoL) assessment — Quality of Life Questionnaire C-30 (QLQ-C30), Impact on Participation and Autonomy Questionnaire (IPAQ) and Musculoskeletal Tumor Society Score (MSTS)
  Arms: Bone or soft tissue sarcoma of the lower extremity; Soft tissue sarcoma of the thigh

SUMMARY:
Primary bone and soft tissue sarcomas are an exceptionally rare form of cancer, collectively accounting for only 1% of all malignancies diagnosed. Sarcomas often occur in the patients' extremities and treatment typically involves limb salvage surgery with bone and/or muscle resection. These surgeries often leave the patients with disfigurements, psychological trauma, and functional disabilities. Perhaps, the most difficult and life-altering decision that patients (and their parents) with primary bone sarcomas about the knee joint have to make, involves choosing the type of surgical procedure that will provide them with the outcome that meets their functional as well as aesthetic expectations.

In literature, the quality of life for patients with osteosarcoma around the knee joint after three different surgical procedures, that is, amputation, endoprosthetic reconstruction and rotationplasty was evaluated. There was found that patients treated with rotationplasty showed significantly higher functional scores compared to the two other groups of patients. Also, researchers investigated the long-term quality of life after bone sarcoma surgery around the knee joint and found that, despite the functional disability, survivors were busy with work, study, relationships, and sometimes they have founded a family.

Most published reports in the literature on assessment of gait in the lower-extremity sarcoma survivors were focused on bone sarcoma patients after wide resection and endoprosthetic reconstruction. To the knowledge of the investigator, there has been no published studies on gait analysis after resection of soft tissue sarcomas (STS) of the lower extremity. The rare and heterogeneous aspects of STS and the paucity of knowledge of movement strategies in these patients hinder the development of effective rehabilitation protocols for recovering movement after resection of STS in the lower limb.

DETAILED DESCRIPTION:
Primary bone and soft tissue sarcomas are an exceptionally rare form of cancer, collectively accounting for only 1% of all malignancies diagnosed. There have been dramatic improvements in the survival rate of sarcoma patients in the past 40 years owing to increasing effectiveness of chemotherapy. This, along with developments in imaging techniques, have led to earlier diagnosis and more accurate preoperative staging. It is estimated that there are nearly 50,000 survivors of bone and soft tissue sarcomas in the United States. 70% of those are younger than the age of 50 years. Whilst traditional treatment for bone tumors used to be amputation, advances in surgical techniques have made limb-salvage procedures a valid alternative method of treatment in 80-85% of patients with primary bone sarcomas.

Sarcomas often occur in the patients' extremities and treatment typically involves limb salvage surgery with bone and/or muscle resection. These surgeries often leave the patients with disfigurements, psychological trauma, and functional disabilities. Perhaps, the most difficult and life-altering decision that patients (and their parents) with primary bone sarcomas about the knee joint have to make, involves choosing the type of surgical procedure that will provide them with the outcome that meets their functional as well as aesthetic expectations. In literature, the quality of life for patients with osteosarcoma around the knee joint after three different surgical procedures, that is, amputation, endoprosthetic reconstruction and rotationplasty was evaluated. There was found that patients treated with rotationplasty showed significantly higher functional scores compared to the two other groups of patients. Also, researchers investigated the long-term quality of life after bone sarcoma surgery around the knee joint and found that, despite the functional disability, survivors were busy with work, study, relationships, and sometimes they have founded a family.

There are few reports available in the literature on the quality of life in sarcoma survivors. It was found that elderly patients, retired patients, and those who live alone need more intensive psychological care. Female patients were found to cope poorly with their disease compared to male gender. It was also found that the physical status greatly influences the overall outcome and quality of life in this group of patients. This stresses the importance of enrolment in tailored rehabilitation programs.

Most published reports in the literature on assessment of gait in the lower-extremity sarcoma survivors were focused on bone sarcoma patients after wide resection and endoprosthetic reconstruction. In literature, the gait pattern after endoprosthetic replacement around the knee joint was studied and found that, despite decreased walking velocity, stride length, and stance phase of the operated limb, these patients still have a symmetrical gait. Also in another report, an electromyographic assessment of gait after bone sarcoma surgery about the knee showed prolonged activation of rectus femoris and hamstring muscles in the affected limb compared to a control group. Other researchers found that limb-salvage patients often adopt a "stiff-legged" gait pattern. These findings are of utmost importance for the development of efficient rehabilitation programs for these patients.

To the knowledge of the investigator, there has been no published studies on gait analysis after resection of soft tissue sarcomas (STS) of the lower extremity. The rare and heterogeneous aspects of STS and the paucity of knowledge of movement strategies in these patients hinder the development of effective rehabilitation protocols for recovering movement after resection of STS in the lower limb. Researchers investigated the knee extension strength and postoperative functional outcome after quadriceps resection for soft tissue sarcoma of the thigh. They found that knee extension strength decreased when the number of resected quadriceps increased and this was associated with lower functional scores. They concluded that good functional results can be expected if at least two quadriceps muscles are preserved. However, no detailed assessment of gait in this group of patients has been published.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent limb salvage surgery for bone or soft tissue sarcoma of the lower extremity at UZ Leuven
* 18 to 95 years old
* Patients should be at least one year post surgery
* Informed consent has obtained

Exclusion Criteria:

* Patients who received major prior surgery of the lower limbs or with any pathology, injury or disorder known to affect the locomotor system
* Skeletally immature individuals
* No informed consent has obtained

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Tumor Society Score (MSTS) | Within a period of 1 year
  To determine the physical and mental health for patients with extremity sarcoma
Quality of Life Questionnaire C-30 (QLQ-C30) | Within a period of 1 year
  To measure cancer patients' physical, psychological and social functions
Participation and Autonomy Questionnaire Questionnaire (IPAQ) | Within a period of 1 year
  To measure health-related physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Wafa, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No